CLINICAL TRIAL: NCT04302727
Title: Randomized Explanatory Trial of a Mediterranean Dietary Pattern Weight Loss Intervention for Primary Care Practices
Brief Title: Delicious Eating for Life in Southern Homes
Acronym: DELISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1712; 1R61HL142680-01A1 (NIH); 4R33HL142680-02 (NIH); 5R33HL142680-03 (NIH)
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-06

CONDITIONS: Weight Loss; Diet, Healthy; Cardiovascular Risk Factor
Keywords: Behavioral weight loss; Mediterranean dietary pattern; Lifestyle program; Inflammatory markers
MeSH Terms: conditions — Weight Loss | interventions — Weight Reduction Programs

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either the intervention group (Med-Diet Weight Loss Program) or an enhanced usual care control group (WW); both groups will participate in the respective programs for two years.
Who Masked: Outcomes Assessor
Masking Description: The investigators (excluding bio-statistician) will be masked to weight change and other major outcomes (will not have access to the data) until all data are collected. The bio-statistician will have access to study group assignment as liaison to the Data Safety Monitoring Committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Med-South Weight Loss Intervention (Experimental): The intervention will be delivered in 3 phases over 24 months: Phase I (4 months) provides a foundation for adopting and maintaining a healthful dietary pattern (Med-style, tailored for the southeastern United States); Phase II (8 months) focuses on weight loss; and Phase III (12 months) on maintenance of or continued weight loss, as appropriate.
  Interventions: Behavioral: Med-South Weight Loss Intervention
- Augmented Usual Care (WW) (Active Comparator): The intervention that will be offered to control group participants is WW™ (formerly known as Weight Watchers). The study will provide access to the 'Workshop + Digital' option of WW™ during the 2 year intervention.
  Interventions: Behavioral: WW

INTERVENTIONS:
Behavioral: Med-South Weight Loss Intervention — Phase I is a 4-month lifestyle program focused on the basics of healthy eating. Phase II (8 months) focuses on weight loss, followed by a year-long (Phase III) focused on weight loss maintenance. In Phase I, the main counseling sessions happen at monthly visits, with added check-in phone calls. In Phase II, the main counseling sessions will occur weekly for 6-8 weeks. There are also check-in phone calls - number based on weight loss progress. During Phase III, there are 2 main visits and follow-up phone calls. Counseling visits will be in-person with a health counselor and by phone. Of the 14 core counseling sessions, the in-person format will be required for only 4 (the 1st session of each Phase and after 2 months of the weight loss program). The program also includes brief phone calls to check on progress towards goals for lifestyle change. The number of phone calls will depend on success in meeting personal weight loss goals in Phase II or keeping the weight off in Phase III.
  Other Names: Delicious Eating for Life in Southern Homes (DELISH) Weight Loss Program
  Arms: Med-South Weight Loss Intervention
Behavioral: WW — If participants are randomized to WW™, they will have access to both the workshop and digital components of the WW™ program for 2 years. The workshop component includes the option of attending weekly group meeting at a WW™ studio (local WW™ office). The digital component can be accessed using the WW™ website or the smart phone App. The study research staff will provide basic instructions on how to use the WW™ digital resources.
  Other Names: Weight Watchers
  Arms: Augmented Usual Care (WW)

SUMMARY:
This study will compare a new weight loss program that focuses on a healthy eating pattern, with WW™ (formally Weight Watchers), an effective and widely available weight loss program. Study researchers have developed an adapted version of the Mediterranean eating pattern to be more acceptable and realistic for southerners; this adapted version is known as "Med-South." Those who take part in the study will be randomly assigned to either the Med-South weight loss program or WW™. Both programs will last for 2 years with measurement visits at the start of the study and at 4-, 12- and 24-month follow-up. While the primary outcome measured by the trial will be weight loss at 24 months, researchers will collect other data which may show additional health benefits of the Med-South diet. The study team will measure blood markers of inflammation, which are known to improve with better diet quality. Researchers will also measure participants' skin carotenoid levels, which increase with greater fruit and vegetable consumption. The study will be conducted within 2 regional catchment areas (n=360 participants) representing a diverse spectrum of patients and settings. Patients with a BMI ≥ 30 kg/m^2 will be enrolled and randomized to intervention or augmented usual care. To assure adequate subgroup representation, ≥ 40% of the sample will have diabetes, ≥ 40% will be male, and ≥ 40% will be African American. The intervention will be delivered in 3 phases over 24 months by research staff: Phase I (4 months) focuses on adopting a Med-style dietary pattern; Phase II (8 months) on weight loss; and Phase III (12 months) on weight loss maintenance. Outcomes will be assessed at 4, 12, and 24 months. The primary outcome is weight loss at 24 months. Secondary outcomes include change in physiologic, behavioral, and psychosocial measures. Researchers will also assess implementation cost and the incremental cost-effectiveness of the intervention relative to the augmented usual care group.

DETAILED DESCRIPTION:
Below, each of the treatment arms is described in detail.

Med-South Weight Loss Program

Most weight loss programs offer weekly one-on-one or group counseling sessions for 16-20 weeks. The Med-South Weight Loss Program is different and is given in 3 phases. The program begins with Phase I, a 4-month lifestyle phase that focuses on the "basics" of healthy eating rather than weight loss. Over the next 8 months in Phase II, we focus on weight loss, followed by a year-long (Phase III) phase to help maintain weight loss. In Phase I, the main counseling sessions happen at monthly visits, to which check-in phone calls are added. In Phase II, the main counseling sessions will occur weekly for 6-8 weeks, depending on participants' progress. There are also check in phone calls-the number will vary based on progress. During Phase III, there are 2 main visits and follow-up phone calls. More details about these visits are in the table below.

Some of the counseling visits will be face-to-face with the counselor and some by phone. Only one member of a family may join this study, but other family members are invited to take part in face-to-face and phone counseling sessions. (As of June 2020, due to COVID-19 only one other family member or friend may come with you to in-person visits.) Of the 14 core counseling sessions), the face-to-face format will be required for only 5 (the 1st session of each Phase, after 2 months of the weight loss program, and approximately 1/2 through the year long maintenance phase). (As of June 2020, due to COVID-19, only these visits will be in person. All the others will be by phone or videoconferencing, until further notice based on updated COVID-19 guidelines.) During face-to-face sessions, the participant and the counselor will sit side-by-side and use a web-based program or the paper format to review educational materials, select dietary goals, and list first steps to reach these goals. (As of June 2020, due to COVID-19, counselor and participant will sit more than 6 feet apart and a large wall mounted monitor will be used to review study materials. This protocol will be followed until further notice based on updated COVID-19 guidelines.) If the phone format is used for major counseling sessions, the participant may view the educational content online or use the paper version. The program also includes brief telephone calls to check on progress towards goals selected at previous sessions and provide support for lifestyle change. The number of phone calls will depend on the participant meeting his/her personal weight loss goals in Phase II or keeping the weight off in Phase III. Detail for each Phase is given below.

Phase I

* 8 total contacts

  * 4 core sessions: the first must be in-person; choice of in-person or phone for all others
  * 4 follow-up phone calls
* Core session = 45-60 min.
* Follow-up call = 15 min.
* total time: 4 - 5 hours

Phase II

* 14 core sessions: the first and third must be in-person; choice of in-person or phone for all others.
* 6-12 follow-up phone calls
* Core session (In-person) = 45-60 min.
* Core session (phone) = 30-45 min.
* Follow-up call = 20-30 min. Total time 8.7 - 14 hours (core) 4.7 - 9.5 hours (Follow-up)

Phase III

* 2 core sessions (both in-person)
* 12-24 follow-up phone calls (1-2 per month)
* Core session (In-person) = 45-60 min.
* Follow-up call = 15-20 min. Total time 1.25 - 2 hours (Core) 3 - 8 hours (Follow-up)

  2-Year Program TOTAL 44 - 60 Contacts -- 21.7 - 38.5 hours

WW™ Weight Loss Program

Those randomized to WW™ will have access to both the Workshop and Digital components of the WW™ program for 2 years. WW offers in-person coaching and community-based learning through weekly Workshops at WW Studios.The Workshop component allows for attending weekly group meeting at a WW™ studio (local WW™ office). (As of June 2020, due to COVID-19, the workshop component will be available in a virtual videoconferencing [Zoom™] format until further notice based on updated COVID-19 guidelines.)

The Digital component can be accessed using the WW™ website or the smart phone App. The digital tools available thought the WW Digital program include food tracking (either manually or with bar code scanning), progress charts, lifestyle coaching with 24/7 chat with a WW Coach, ability to track activity (manually or by syncing a fitness tracking device), incentives for behavior change (WellnessWins), recipes, and even local restaurant recommendations using GPS. Those in the WW group will also have access to Connect, WW's members-only digital community.

The WW™ program uses "SmartPoints" assigned to foods based on energy content and nutritional value, allocating a certain number of points to users daily based on their starting weight, weight loss goals, age and sex. Participants will receive a personalized SmartPoints budget made up of Daily SmartPoints, plus some extra Weekly SmartPoints for those days when a cushion is needed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* English speaking
* Ages 18-75 (inclusive)
* BMI > or = 30 kg/m^2
* Approval for participation by primary care clinician
* Established patient at participating practice defined as at least one prior visit at the practice within the prior 2 years
* Access to telephone
* No plans to move from the area for at least 1 year
* Free living to the extent that participant has control over dietary intake
* Those with known cardiovascular disease will be allowed to participant

Exclusion Criteria:

* Participant in intensive weight loss program (more than 6 visits) in the prior year
* Another family member or household member is a study participant. Only one member of each household may take part in this study.
* Considering bariatric surgery in the next year or prior bariatric surgery
* Type 1 diabetes. Rationale is patients with type 1 diabetes already received intensive dietary counseling with a focus on total and distribution of daily carbohydrates.
* Pregnancy/breastfeeding or intended pregnancy in the next year
* History of malignancy, other than non-melanoma skin cancer, unless surgically or medically cured > 5 years ago or in remission. Patients with localized prostate and breast cancer diagnosed during the course of routine screening will not be excluded.
* Advanced kidney disease (estimated creatinine clearance < 30 mL/min)
* Known drug or alcohol misuse in the past 2 years
* Known psychosis or major psychiatric illness. Those with major depression who have responded to treatment may participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen D Samuel-Hodge, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Thomas C Keyserling, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center for Health Promotion and Disease Prevention, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: Approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Keyserling TC, Samuel-Hodge CD, Pitts SJ, Garcia BA, Johnston LF, Gizlice Z, Miller CL, Braxton DF, Evenson KR, Smith JC, Davis GB, Quenum EL, Elliott NT, Gross MD, Donahue KE, Halladay JR, Ammerman AS. A community-based lifestyle and weight loss intervention promoting a Mediterranean-style diet pattern evaluated in the stroke belt of North Carolina: the Heart Healthy Lenoir Project. BMC Public Health. 2016 Aug 5;16:732. doi: 10.1186/s12889-016-3370-9. PMID 27495295
- [Background] Keyserling TC, Samuel Hodge CD, Jilcott SB, Johnston LF, Garcia BA, Gizlice Z, Gross MD, Savinon CE, Bangdiwala SI, Will JC, Farris RP, Trost S, Ammerman AS. Randomized trial of a clinic-based, community-supported, lifestyle intervention to improve physical activity and diet: the North Carolina enhanced WISEWOMAN project. Prev Med. 2008 Jun;46(6):499-510. doi: 10.1016/j.ypmed.2008.02.011. Epub 2008 Feb 15. PMID 18394692
- [Background] Keyserling TC, Sheridan SL, Draeger LB, Finkelstein EA, Gizlice Z, Kruger E, Johnston LF, Sloane PD, Samuel-Hodge C, Evenson KR, Gross MD, Donahue KE, Pignone MP, Vu MB, Steinbacher EA, Weiner BJ, Bangdiwala SI, Ammerman AS. A comparison of live counseling with a web-based lifestyle and medication intervention to reduce coronary heart disease risk: a randomized clinical trial. JAMA Intern Med. 2014 Jul;174(7):1144-57. doi: 10.1001/jamainternmed.2014.1984. PMID 24861959
- [Background] Embree GG, Samuel-Hodge CD, Johnston LF, Garcia BA, Gizlice Z, Evenson KR, DeWalt DA, Ammerman AS, Keyserling TC. Successful long-term weight loss among participants with diabetes receiving an intervention promoting an adapted Mediterranean-style dietary pattern: the Heart Healthy Lenoir Project. BMJ Open Diabetes Res Care. 2017 Mar 29;5(1):e000339. doi: 10.1136/bmjdrc-2016-000339. eCollection 2017. PMID 28405344
- [Background] Samuel-Hodge CD, Holder-Cooper JC, Gizlice Z, Davis G, Steele SP, Keyserling TC, Kumanyika SK, Brantley PJ, Svetkey LP. Family PArtners in Lifestyle Support (PALS): Family-based weight loss for African American adults with type 2 diabetes. Obesity (Silver Spring). 2017 Jan;25(1):45-55. doi: 10.1002/oby.21700. Epub 2016 Dec 2. PMID 27911049
- [Background] Samuel-Hodge CD, Garcia BA, Johnston LF, Gizlice Z, Ni A, Cai J, Kraschnewski JL, Gustafson AA, Norwood AF, Glasgow RE, Gold AD, Graham JW, Evenson KR, Trost S, Keyserling TC. Translation of a behavioral weight loss intervention for mid-life, low-income women in local health departments. Obesity (Silver Spring). 2013 Sep;21(9):1764-73. doi: 10.1002/oby.20317. Epub 2013 May 24. PMID 23408464
- [Background] Samuel-Hodge CD, Johnston LF, Gizlice Z, Garcia BA, Lindsley SC, Bramble KP, Hardy TE, Ammerman AS, Poindexter PA, Will JC, Keyserling TC. Randomized trial of a behavioral weight loss intervention for low-income women: the Weight Wise Program. Obesity (Silver Spring). 2009 Oct;17(10):1891-9. doi: 10.1038/oby.2009.128. Epub 2009 Apr 30. PMID 19407810
- [Derived] Saraiya VM, Berkowitz SA, Johnston LF, Couper DJ, Sotres-Alvarez D, Lyons KM, Thaxton CK, Skinner HG, Samuel-Hodge CD, Keyserling TC. An Evaluation of Primary Care Clinician Referrals for Behavioral Weight Loss Counseling. J Prim Care Community Health. 2024 Jan-Dec;15:21501319241308054. doi: 10.1177/21501319241308054. PMID 39690977

RESULTS

PARTICIPANT FLOW:
Groups:
- Augmented Usual Care (WW): The intervention that will be offered to control group participants is WW™ (also known as Weight Watchers). The study will provide access to the 'Workshop + Digital' option of WW™ during the 2 year intervention.
  WW: If participants are randomized to WW™, they will have access to both the workshop and digital components of the WW™ program for 2 years. The workshop component includes the option of attending weekly group meeting at a WW™ studio (local WW™ office). The digital component can be accessed using the WW™ website or the smart phone App. The study research staff will provide basic instructions on how to use the WW™ digital resources.
Period: Overall Study
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Started | 182 | 178
Completed | 118 | 129
Not Completed | 64 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW) | Total
Number analyzed (Participants) | 182 | 178 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.5) | 55.0 (11.6) | 54.7 (12.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 78 | 80 | 158
  Female | 104 | 96 | 200
  Non-Binary | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 176 | 166 | 342
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 55 | 64 | 119
  White | 113 | 102 | 215
  More than one race | 9 | 7 | 16
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 182 | 178 | 360

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change From Baseline to Month 24
Description: Weight will be collected by study staff who are masked to treatment using scales tested monthly for accuracy up to 350 pounds.
Time Frame: Baseline, Month 24
Measure: Mean (Standard Deviation); unit: percentage weight change
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 118 | 129
percentage weight change | -4.4 (7.45) | -3.8 (6.00)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Test type: Superiority; p = 0.43, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Fully adjusted model; Test type: Superiority; p = 0.64, Mixed Models Analysis; Median Difference (Net) = 0.37, 95% CI 2-sided [-1.19 to 1.93]

2. Secondary Outcome: Percent Weight Change From Baseline to Months 4 and 12
Description: as for outcome 1
Time Frame: Baseline, Months 4 and 12
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: percentage weight change
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 146 | 152
percentage weight change
  Baseline, Month 4 | -0.9 (3.96) | -4.4 (5.01)
  Baseline, Month 12: number analyzed (Participants) | 112 | 121
  Baseline, Month 12 | -4.6 (6.20) | -4.3 (6.18)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.67, t-test, 2 sided

3. Secondary Outcome: Percentage Weight From Baseline Through Follow-Up by Sub-Groups
Description: Weight will be collected by study staff who are masked to treatment using scales tested monthly for accuracy up to 350 pounds. Assess difference between study groups in percentage losing ≥ 5% body weight for all participants and across 3 pre-specified subgroups: 1) participants with vs. without diabetes; 2) females vs. males; and 3) Whites vs. African Americans.
Time Frame: Baseline, Months 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: percentage weight change
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 146 | 152
percentage weight change
  Participants with diabetes-Baseline, Month 4: number analyzed (Participants) | 42 | 49
  Participants with diabetes-Baseline, Month 4 | -1.7 (3.63) | -3.7 (4.56)
  Participants without diabetes-Baseline, Month 4: number analyzed (Participants) | 104 | 103
  Participants without diabetes-Baseline, Month 4 | -0.6 (4.06) | -4.7 (5.19)
  Females-Baseline, Month 4: number analyzed (Participants) | 83 | 85
  Females-Baseline, Month 4 | -0.3 (3.77) | -4.0 (4.77)
  Males-Baseline, Month 4: number analyzed (Participants) | 63 | 67
  Males-Baseline, Month 4 | -1.7 (4.08) | -4.8 (5.29)
  Whites-Baseline, Month 4: number analyzed (Participants) | 100 | 92
  Whites-Baseline, Month 4 | -1.2 (3.96) | -5.6 (5.38)
  African Americans-Baseline, Month 4: number analyzed (Participants) | 46 | 60
  African Americans-Baseline, Month 4 | -0.5 (3.95) | -2.5 (3.68)
  Participants with diabetes-Baseline, Month 12: number analyzed (Participants) | 34 | 42
  Participants with diabetes-Baseline, Month 12 | -4.2 (5.97) | -3.9 (6.78)
  Participants without diabetes-Baseline, Month 12: number analyzed (Participants) | 78 | 79
  Participants without diabetes-Baseline, Month 12 | -4.8 (6.32) | -4.5 (5.87)
  Females-Baseline, Month 12: number analyzed (Participants) | 61 | 71
  Females-Baseline, Month 12 | -3.3 (6.04) | -3.7 (5.98)
  Males-Baseline, Month 12: number analyzed (Participants) | 51 | 50
  Males-Baseline, Month 12 | -6.2 (6.06) | -5.0 (6.44)
  Whites-Baseline, Month 12: number analyzed (Participants) | 77 | 70
  Whites-Baseline, Month 12 | -5.4 (6.85) | -5.6 (6.53)
  African Americans-Baseline, Month 12: number analyzed (Participants) | 35 | 51
  African Americans-Baseline, Month 12 | -3.0 (4.09) | -2.5 (5.19)
  Participants with diabetes-Baseline, Month 24: number analyzed (Participants) | 38 | 45
  Participants with diabetes-Baseline, Month 24 | -4.7 (6.57) | -5.0 (6.30)
  Participants without diabetes-Baseline, Month 24: number analyzed (Participants) | 80 | 84
  Participants without diabetes-Baseline, Month 24 | -4.3 (7.87) | -3.1 (5.78)
  Females-Baseline, Month 24: number analyzed (Participants) | 64 | 70
  Females-Baseline, Month 24 | -3.6 (7.69) | -3.6 (6.40)
  Males-Baseline, Month 24: number analyzed (Participants) | 54 | 59
  Males-Baseline, Month 24 | -5.5 (7.08) | -3.9 (5.54)
  Whites-Baseline, Month 24: number analyzed (Participants) | 80 | 76
  Whites-Baseline, Month 24 | -4.9 (7.73) | -4.2 (5.99)
  African Americans-Baseline, Month 24: number analyzed (Participants) | 38 | 53
  African Americans-Baseline, Month 24 | -3.5 (6.81) | -3.1 (6.02)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Participants with diabetes-Month 4; Test type: Superiority; p = 0.02, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Participants without diabetes-Month 4; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Participants with diabetes-Month 12; Test type: Superiority; p = 0.82, t-test, 2 sided
Statistical Analysis 4: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Participants without diabetes-Month 12; Test type: Superiority; p = 0.75, t-test, 2 sided
Statistical Analysis 5: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Participants with diabetes-Month 24; Test type: Superiority; p = 0.87, t-test, 2 sided
Statistical Analysis 6: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Participants without diabetes-Month 24; Test type: Superiority; p = 0.27, t-test, 2 sided
Statistical Analysis 7: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Females-Month 4; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Females-Month 12; Test type: Superiority; p = 0.66, t-test, 2 sided
Statistical Analysis 9: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Females-Month 24; Test type: Superiority; p = 0.96, t-test, 2 sided
Statistical Analysis 10: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Males-Month 4; Test type: Superiority; p = 0.0003, t-test, 2 sided
Statistical Analysis 11: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Males-Month 12; Test type: Superiority; p = 0.34, t-test, 2 sided
Statistical Analysis 12: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Males-Month 24; Test type: Superiority; p = 0.20, t-test, 2 sided
Statistical Analysis 13: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Whites-Month 4; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 14: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Whites-Month 12; Test type: Superiority; p = 0.83, t-test, 2 sided
Statistical Analysis 15: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Whites-Month 24; Test type: Superiority; p = 0.54, t-test, 2 sided
Statistical Analysis 16: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); African Americans-Month 4; Test type: Superiority; p = 0.008, t-test, 2 sided
Statistical Analysis 17: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); African Americans-Month 12; Test type: Superiority; p = 0.58, t-test, 2 sided
Statistical Analysis 18: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); African Americans-Month 24; Test type: Superiority; p = 0.79, t-test, 2 sided

4. Secondary Outcome: Mean Weight Change From Baseline Through Follow-Up
Description: Weight will be collected by study staff who are masked to treatment.
Time Frame: Baseline, Months 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 146 | 152
Kg
  Baseline, Month 4 | -1.1 (4.38) | -4.8 (5.60)
  Baseline, Month 12: number analyzed (Participants) | 112 | 121
  Baseline, Month 12 | -5.1 (6.85) | -4.6 (6.81)
  Baseline, Month 24: number analyzed (Participants) | 118 | 129
  Baseline, Month 24 | -5.1 (8.57) | -4.1 (6.36)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.57, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.32, t-test, 2 sided

5. Secondary Outcome: Mean Change in Systolic Blood Pressure From Baseline Through Follow-Up
Description: Blood pressure assessed by Omron-907xl, average of 3 readings.
Time Frame: Baseline, Months 4, 12, and 24
Population: Blood pressure assessed by Omron-907xl if an average of 3 error-free readings were obtained.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 142 | 152
mm Hg
  Baseline, Month 4 | -4.1 (12.37) | -4.5 (12.17)
  Baseline, Month 12: number analyzed (Participants) | 110 | 121
  Baseline, Month 12 | -6.5 (13.62) | -5.2 (13.14)
  Baseline, Month 24: number analyzed (Participants) | 115 | 127
  Baseline, Month 24 | -4.7 (14.23) | -3.9 (14.23)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.77, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.48, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.68, t-test, 2 sided

6. Secondary Outcome: Mean Change in Diastolic Blood Pressure From Baseline Through Follow-Up
Description: Blood pressure assessed by Omron-907xl, average of 3 readings.
Time Frame: Baseline, Months 4, 12, and 24
Population: Blood pressure assessed by Omron-907xl if an average of 3 error-free readings were obtained.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 142 | 151
mm Hg
  Baseline, Month 4 | -3.4 (7.78) | -3.3 (7.72)
  Baseline, Month 12: number analyzed (Participants) | 110 | 121
  Baseline, Month 12 | -4.6 (8.74) | -3.9 (7.62)
  Baseline, Month 24: number analyzed (Participants) | 115 | 127
  Baseline, Month 24 | -3.2 (8.93) | -3.2 (9.24)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.91, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.52, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.97, t-test, 2 sided

7. Secondary Outcome: Mean Change in Total Cholesterol From Baseline Through Follow-Up
Description: Total cholesterol assessed by commercial lab (LabCorp).
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants with successful phlebotomy.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 140 | 142
mg/dL
  Baseline, Month 4 | -1.4 (24.34) | -4.3 (22.47)
  Baseline, Month 12: number analyzed (Participants) | 107 | 108
  Baseline, Month 12 | -5.1 (29.86) | -3.6 (28.43)
  Baseline, Month 24: number analyzed (Participants) | 111 | 115
  Baseline, Month 24 | -2.6 (31.89) | -10.2 (35.32)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.29, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Test type: Superiority; p = 0.71, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.09, t-test, 2 sided

8. Secondary Outcome: Mean Change in HDL-Cholesterol From Baseline Through Follow-Up
Description: HDL-Cholesterol assessed by commercial lab (LabCorp).
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants with successful phlebotomy.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 140 | 142
mg/dL
  Baseline, Month 4 | -0.1 (6.16) | -0.1 (6.60)
  Baseline, Month 12: number analyzed (Participants) | 107 | 108
  Baseline, Month 12 | 1.7 (7.42) | 1.4 (3.73)
  Baseline, Month 24: number analyzed (Participants) | 111 | 115
  Baseline, Month 24 | 3.0 (8.43) | 2.9 (7.43)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.96, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.77, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.94, t-test, 2 sided

9. Secondary Outcome: Mean Change in Triglycerides From Baseline Through Follow-Up
Description: Triglycerides as assessed by commercial lab (LabCorp).
Time Frame: Baseline, Month 4, 12, and 24
Population: Participants with successful phlebotomy who reported fasting.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 125 | 123
mg/dL
  Baseline, Month 4 | -6.1 (52.6) | -9.4 (34.40)
  Baseline, Month 12: number analyzed (Participants) | 96 | 93
  Baseline, Month 12 | -8.6 (115.9) | -5.8 (44.30)
  Baseline, Month 24: number analyzed (Participants) | 96 | 106
  Baseline, Month 24 | -10.4 (64.07) | -4.2 (48.09)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.55, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.83, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.44, t-test, 2 sided

10. Secondary Outcome: Mean Change LDL-cholesterol From Baseline Through Follow-up
Description: Calculated from above lipid assessments by commercial lab (LabCorp).
Time Frame: Baseline, Month 4, 12, and 24
Population: Participants with successful phlebotomy who reported fasting.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 124 | 123
mg/dL
  Baseline, Month 4 | -1.7 (20.81) | -2.6 (21.98)
  Baseline, Month 12: number analyzed (Participants) | 95 | 83
  Baseline, Month 12 | -5.59 (21.80) | -4.97 (25.84)
  Baseline, Month 24: number analyzed (Participants) | 96 | 106
  Baseline, Month 24 | -5.87 (24.47) | -13.90 (31.25)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.99, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.71, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.44, t-test, 2 sided

11. Secondary Outcome: Mean Change in A1c From Baseline Through Follow-Up
Description: A1c assessed by commercial lab (LabCorp).
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants with successful phlebotomy.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 138 | 141
percent
  Baseline, Month 4 | 0.0 (0.62) | -0.2 (0.54)
  Baseline, Month 12: number analyzed (Participants) | 105 | 108
  Baseline, Month 12 | -0.1 (0.58) | -0.2 (0.75)
  Baseline, Month 24: number analyzed (Participants) | 109 | 114
  Baseline, Month 24 | 0.0 (0.60) | -0.2 (0.80)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.42, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.02, t-test, 2 sided

12. Secondary Outcome: Mean Change in CRP (C-Reactive Protein) From Baseline Through Follow-Up
Description: CRP assessed by commercial lab (LabCorp).
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants with successful phlebotomy.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 139 | 143
mg/L
  Baseline, Month 4 | 0.1 (2.61) | -0.6 (4.72)
  Baseline, Month 12: number analyzed (Participants) | 107 | 108
  Baseline, Month 12 | 1.0 (5.27) | 0.4 (8.28)
  Baseline, Month 24: number analyzed (Participants) | 110 | 115
  Baseline, Month 24 | -0.7 (3.22) | -1.1 (5.30)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.10, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.56, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Test type: Superiority; p = 0.50, t-test, 2 sided

13. Secondary Outcome: Mean Change in Interleukin (IL) IL-6 From Baseline Through Follow-Up
Description: Assessed by independent lab blinded to participant arm.
Time Frame: Baseline, Month 4, 12, and 24
Population: Participants with successful phlebotomy who reported fasting and who had a measurable level.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 126 | 126
pg/mL
  Baseline, Month 4 | -0.63 (4.21) | -0.35 (3.30)
  Baseline, Month 12: number analyzed (Participants) | 97 | 96
  Baseline, Month 12 | -0.64 (4.90) | -0.14 (5.55)
  Baseline, Month 24: number analyzed (Participants) | 82 | 94
  Baseline, Month 24 | -0.20 (3.37) | -1.60 (3.82)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4, comparison performed on log base 2 transformation of fluorescence data; Test type: Superiority; p = 0.96, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12, comparison performed on log base 2 transformation of fluorescence data; Test type: Superiority; p = 0.88, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24, comparison performed on log base 2 transformation of fluorescence data; Test type: Superiority; p = 0.29, t-test, 2 sided

14. Secondary Outcome: Mean Change in Tumor Necrosis Factor (TNF) TNF-alpha From Baseline Through Follow-Up
Description: Assessed by independent lab blinded to participant arm.
Time Frame: Baseline, Month 4, 12, and 24
Population: Participants with successful phlebotomy who reported fasting and who had a measurable level. The numbers differ from IL-6 due to number of participants with results below the lower limit of the assay.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 128 | 129
pg/mL
  Baseline, Month 4 | -0.39 (6.87) | -0.03 (3.20)
  Baseline, Month 12: number analyzed (Participants) | 98 | 101
  Baseline, Month 12 | -0.69 (10.52) | -0.30 (3.14)
  Baseline, Month 24: number analyzed (Participants) | 95 | 107
  Baseline, Month 24 | -1.27 (10.94) | -0.16 (3.25)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4, comparison performed on log base 2 transformation of fluorescence data; Test type: Superiority; p = 0.82, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12, comparison performed on log base 2 transformation of fluorescence data; Test type: Superiority; p = 0.25, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24, comparison performed on log base 2 transformation of fluorescence data; Test type: Superiority; p = 0.48, t-test, 2 sided

15. Secondary Outcome: Mean Change in Skin Carotenoids From Baseline Through Follow-Up
Description: Evaluated as the sum of 3 measures assessed by veggie-meter by Longevity Link Corporation. The Veggie Meter produces a score from 0 to 800, with higher scores indicating greater skin carotenoid levels, which suggest a greater intake of fruits and vegetables.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 143 | 152
score on a scale
  Baseline, Month 4 | 8.5 (50.23) | 31.8 (66.43)
  Baseline, Month 12: number analyzed (Participants) | 112 | 121
  Baseline, Month 12 | 24.3 (69.87) | 30.8 (81.07)
  Baseline, Month 24: number analyzed (Participants) | 117 | 127
  Baseline, Month 24 | 13.5 (62.67) | 12.6 (70.85)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.0007, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.51, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.91, t-test, 2 sided

16. Secondary Outcome: Mean Change in Quality of Life Scale From Baseline Through Follow-Up
Description: The Euro Quality of Life Three Dimensions Questionnaire EQ-5D-3L ( EuroQol five-dimensional three-level questionnaire) scale measures patients' quality of healthy living. It has 5 items (Mobility, Self-care, Usual activities, Pain/discomfort, Depression/anxiety). Each item contains 3 levels: 1=no problems; 2=some problems; 3=extreme problems. The higher the score has the worse the health. Then, the score calculation of the European Five-Dimensional Health Scale is based on the calculation formula published for U.S. populations. Based on 3 combinations of different severity for the 5 items, a score of 0 to 1 is obtained which is called the EQ-5D-3L index and reported here. 0 is the least healthy and 1 is the most healthy.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 140 | 147
score on a scale
  Baseline, Month 4 | 0.009 (0.11) | 0.012 (0.11)
  Baseline, Month 12: number analyzed (Participants) | 109 | 113
  Baseline, Month 12 | 0.005 (0.12) | 0.012 (0.13)
  Baseline, Month 24: number analyzed (Participants) | 107 | 118
  Baseline, Month 24 | -0.009 (0.16) | 0.000 (0.13)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.83, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.68, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.64, t-test, 2 sided

17. Secondary Outcome: Mean Change in Alternate Healthy Eating Index (AHEI)-2010 From Baseline Through Follow-Up
Description: The AHEI-2010 is calculated from items on the Willett Food Frequency Questionnaire. It addresses intake of foods and nutrients consistently associated with lower risk for chronic diseases in the literature. The AHEI-2010 score is comprised of 11 sub-scales, each scored from 0 to 10, yielding a total score with a range of 0-110. A higher score indicates a more healthful dietary pattern.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures, completed the Harvard-Willett Food Frequency Questionnaire, and had plausible daily energy intake. For women this was defined as daily kcal intake between 500 and 3500 kcal inclusive. For men this was defined as daily kcal intake between 800 and 4200 kcal inclusive.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 140 | 147
score on a scale
  Baseline, Month 4 | 8.2 (8.97) | 2.8 (9.67)
  Baseline, Month 12: number analyzed (Participants) | 111 | 113
  Baseline, Month 12 | 8.8 (9.18) | 2.4 (9.51)
  Baseline, Month 24: number analyzed (Participants) | 107 | 118
  Baseline, Month 24 | 6.6 (9.68) | 3.0 (9.35)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.005, t-test, 2 sided

18. Secondary Outcome: Mean Change in Global Physical Activity Questionnaire (GPAQ) From Baseline Through Follow-Up
Description: The GPAQ was developed by the World Health Organization (WHO) for physical activity surveillance. It collects information on physical activity participation in three settings (or domains) as well as sedentary behavior. The domains are: activity at work, travel to and from places, and recreational activities. The summary measure will be the sum of all moderate and vigorous activity per week (measured in hours) for the domains mentioned with a higher score indicating more physical activity.
Time Frame: Baseline, Month 4, 12, and 24
Population: The reduced number at follow-up reflects participants that did not return for the measurement visit and those who did not report any moderate or vigorous activity.
Measure: Median (Inter-Quartile Range); unit: hours/week
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 104 | 114
hours/week
  Baseline, Month 4 | 0.92 [-3.04 to 3.50] | 1.00 [-2.75 to 3.25]
  Baseline, Month 12: number analyzed (Participants) | 85 | 91
  Baseline, Month 12 | 1.67 [-0.67 to 6.33] | 1.00 [-1.83 to 5.50]
  Baseline, Month 24: number analyzed (Participants) | 87 | 88
  Baseline, Month 24 | 0.17 [-4.53 to 6.00] | 0.90 [-2.16 to 5.50]
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Test type: Superiority; p = 0.92, Wilcoxon (Mann-Whitney) — Month 4
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Mean Change in Weight Loss Self-Efficacy From Baseline Through Follow-Up
Description: The Weight Efficacy Lifestyle Questionnaire Short-Form (WEL-SF1) is a short version of the original Weight-Efficacy Lifestyle Questionnaire and includes 8 questions and 1 situational component representing "confidence in ability to resist eating." Three of the questions are related to emotional eating situations, two to availability, one to social pressure, one to positive activities, and one to physical discomfort. Scoring: The instrument range scores on a Likert-scale from 0 (not at all confident) to 10 (very confident), with sum scores between 0 and 80. High scores are associated with high eating self-efficacy.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 141 | 151
score on a scale
  Baseline, Month 4 | 2.9 (14.57) | 1.60 (13.50)
  Baseline, Month 12: number analyzed (Participants) | 110 | 120
  Baseline, Month 12 | 5.0 (14.60) | 0.4 (16.90)
  Baseline, Month 24: number analyzed (Participants) | 111 | 124
  Baseline, Month 24 | 5.3 (16.09) | 2.8 (14.97)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.44, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.28, t-test, 2 sided

20. Secondary Outcome: Mean Change in Dietary Self-Regulation From Baseline Through Follow-Up
Description: Treatment Self-regulation Questionnaire (TSRQ) measures the quality of motivation for a particular health goal. Motivation is psychological energy directed at a particular goal such as weight loss. The autonomous self-regulation sub-scale of the TSRQ was used.This 6-item scale will focus on the reasons why people would either start eating a healthier diet or continue to do so. Scoring: Participants rate each statement on a 7-point Likert scale ranging from 1 (not at all true) to 7 (very true). It assesses the degree to which a person's motivation for eating a healthy diet is autonomous or self-determined. Possible scores range from 6 to 42 wtih higher scores indicating greater motivation.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 141 | 151
score on a scale
  Baseline, Month 4 | 0.1 (0.90) | 0.0 (1.05)
  Baseline, Month 12: number analyzed (Participants) | 110 | 120
  Baseline, Month 12 | 0.2 (0.93) | -0.1 (1.03)
  Baseline, Month 24: number analyzed (Participants) | 111 | 124
  Baseline, Month 24 | 0.1 (1.07) | -0.3 (1.08)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.32, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.005, t-test, 2 sided

21. Secondary Outcome: Mean Change in Eating Attitudes From Baseline Through Follow-Up (Cognitive Restraint)
Description: The Cognitive Restraint subscale of the Three Factor Eating Questionnaire has 6 items and measures one of the three dimensions of eating attitudes. The instrument scoring range for each item is based on a Likert-scale from 1 (definitely false) to 4 (definitely true) with scores ranging from 6 and 24. Higher scores indicate greater cognitive restraint.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 141 | 151
score on a scale
  Baseline, Month 4 | 1.7 (3.34) | 2.3 (3.09)
  Baseline, Month 12: number analyzed (Participants) | 110 | 120
  Baseline, Month 12 | 2.5 (3.75) | 1.6 (3.18)
  Baseline, Month 24: number analyzed (Participants) | 111 | 124
  Baseline, Month 24 | 2.3 (3.79) | 1.8 (2.93)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.10, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.16, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.27, t-test, 2 sided

22. Secondary Outcome: Mean Change in Eating Attitudes From Baseline Through Follow-Up (Uncontrolled Eating)
Description: The uncontrolled eating subscale of the Three Factor Eating Questionnaire has 9 items and measures one of the three dimensions of eating attitudes. The instrument scoring range for each item is based on a Likert-scale from 1 (definitely false) to 4 (definitely true) with scores ranging from 9 and 36. Higher scores indicate greater uncontrolled eating.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 141 | 151
score on a scale
  Baseline, Month 4 | -1.2 (3.40) | -0.5 (3.19)
  Baseline, Month 12: number analyzed (Participants) | 110 | 120
  Baseline, Month 12 | -2.0 (3.87) | -0.8 (3.88)
  Baseline, Month 24: number analyzed (Participants) | 111 | 124
  Baseline, Month 24 | -1.9 (3.76) | -0.1 (3.57)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.10, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.06, t-test, 2 sided

23. Secondary Outcome: Mean Change in Eating Attitudes From Baseline Through Follow-Up (Emotional Eating)
Description: The emotional eating subscale of the Three Factor Eating Questionnaire has 3 items and measures one of the three dimensions of eating attitudes. The instrument scoring range for each item is based on a Likert-scale from 1 (definitely false) to 4 (definitely true) with scores ranging from 3 and 12. Higher scores indicate greater emotional eating.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 141 | 151
score on a scale
  Baseline, Month 4 | -0.4 (7.71) | -0.6 (1.69)
  Baseline, Month 12: number analyzed (Participants) | 110 | 120
  Baseline, Month 12 | -0.6 (1.66) | -0.3 (1.98)
  Baseline, Month 24: number analyzed (Participants) | 111 | 124
  Baseline, Month 24 | -0.6 (1.84) | -0.5 (1.91)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.41, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.24, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.74, t-test, 2 sided

24. Secondary Outcome: Mean Change in Diet Self-Efficacy From Baseline Through Follow-Up
Description: Perceived self-efficacy is regarded as a suitable predictor of reported health behaviors. This 5-item scale of perceived self-efficacy measures self-efficacy related to healthful eating behaviors. Responses are on a 4-point scale of 'very uncertain' to 'very certain.' Total scores range from 5-20 with higher scores indicating higher perceived self-efficacy.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 142 | 151
score on a scale
  Baseline, Month 4 | 0.5 (3.78) | -0.1 (3.28)
  Baseline, Month 12: number analyzed (Participants) | 111 | 120
  Baseline, Month 12 | 0.5 (4.21) | -0.4 (3.51)
  Baseline, Month 24: number analyzed (Participants) | 112 | 124
  Baseline, Month 24 | -0.1 (4.58) | -0.8 (3.58)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.13, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p = 0.10, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p = 0.12, t-test, 2 sided

25. Secondary Outcome: Mean Change in Self-Weighing Behaviors From Baseline Through Follow-Up
Description: EARLY Self-Weighing Questionnaire: This is a 1-item screener measures frequency of self-weighing. It was adapted from the Pound of Prevention Health Habits Questionnaire. Those reporting a higher weighing frequency had greater 24-month weight loss or less weight gain. Scoring: Higher scores indicate higher frequency of self-weighing. Responses are based on a 7-point scale ranging from 1 = never; 2 = once a year or less; 3= every couple of months; 4 = about once a month; 5 = about once a week; 6 = about once a day; and 7 = more than once a day.
Time Frame: Baseline, Month 4, 12, and 24
Population: Data reported for all participants who returned for follow-up measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 141 | 151
score on a scale
  Baseline, Month 4 | 1.1 (1.60) | 0.6 (1.25)
  Baseline, Month 12: number analyzed (Participants) | 110 | 120
  Baseline, Month 12 | 1.7 (1.64) | 0.5 (1.24)
  Baseline, Month 24: number analyzed (Participants) | 111 | 124
  Baseline, Month 24 | 1.5 (1.57) | 0.3 (1.28)
Statistical Analysis 1: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 4; Test type: Superiority; p = 0.002, t-test, 2 sided
Statistical Analysis 2: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 12; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Med-South Weight Loss Intervention vs Augmented Usual Care (WW); Month 24; Test type: Superiority; p < 0.001, t-test, 2 sided

26. Secondary Outcome: Economic Outcome--Incremental Cost-Effectiveness
Description: Computed as the incremental cost per kilogram of weight loss relative to control. The budgetary assessment will quantify the total and per participant costs of intervention delivery from the health system perspective using an Activity Based Costing (ABC) approach and cost tracking forms that the health economist (Finkelstein) has developed and refined in past behavioral trials. Using this approach, all relevant labor, materials and supplies, contracted services, and other relevant costs required to deliver the interventions will be captured by key activities
Time Frame: Month 24
Measure: Number; unit: U.S. dollars/Kg
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 118 | 129
U.S. dollars/Kg | NA — Below the level of detection since the adjusted difference in percent weight change between study arms was minimal. The effectiveness results were equivalent, resulting in a zero denominator in the Incremental Cost-Effectiveness Ratio (ICER) calculation. This made the ICER mathematically undefined, and no participants were analyzed for this outcome | NA — Below the level of detection since the adjusted difference in percent weight change between study arms was minimal. The effectiveness results were equivalent, resulting in a zero denominator in the Incremental Cost-Effectiveness Ratio (ICER) calculation. This made the ICER mathematically undefined, and no participants were analyzed for this outcome

27. Secondary Outcome: Economic Outcome--Incremental Cost Per Quality Adjusted Life Year (QALY) Gained
Description: The numerator for this analysis will be the incremental program delivery costs of the intervention relative to control, minus any cost offsets based on differences in health services and medication use across arms. The denominator will be the incremental QALYs based on average differences in Euro Quality of Life five Dimensions Questionnaire (EQ-5D-5L) scores across arms collected at each assessment point. These scores can be used to quantify net QALY differences during the intervention period.
  EQ-5D-5L scale measures patients' quality of healthy living. It has 5 items (Mobility, Self-care, Usual activities, Pain/discomfort, Depression/anxiety). The score calculation of the European Five-Dimensional Health Scale is based on the calculation formula published by the EuroQol Group. Based on 5 combinations of different severity levels, a score of 0 to 1 is obtained. 0 is the least healthy and 1 is the most healthy.
Time Frame: Month 24
Measure: Number; unit: U.S. dollars per QALY
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
Number analyzed (Participants) | 118 | 129
U.S. dollars per QALY | NA — Below the level of detection since the adjusted difference in percent weight change between study arms was minimal. The effectiveness results were equivalent, resulting in a zero denominator in the Incremental Cost-Effectiveness Ratio (ICER) calculation. This made the ICER mathematically undefined, and no participants were analyzed for this outcome. | NA — Below the level of detection since the adjusted difference in percent weight change between study arms was minimal. The effectiveness results were equivalent, resulting in a zero denominator in the Incremental Cost-Effectiveness Ratio (ICER) calculation. This made the ICER mathematically undefined, and no participants were analyzed for this outcome.

ADVERSE EVENTS:
Time Frame: From the time of randomization to the final follow-up visit, a total of approximately 24 months (the defined window for the final follow-up was 23-30 months). For those who did not attend the final follow-up visit, reports for hospitalization were reviewed from the electronic health record for 2 years post randomization.
Description: Adverse events were captured using the electronic health record report for hospitalizations and by participant-completed surveys at follow-up visits.
Arm/Group | Med-South Weight Loss Intervention | Augmented Usual Care (WW)
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/178
Serious Adverse Events (participants affected / at risk) | 24/182 | 10/178
Other Adverse Events (participants affected / at risk) | 27/182 | 31/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Med-South Weight Loss Intervention (N=182) | Augmented Usual Care (WW) (N=178)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 2 (5) | 0 (0)
Subdural Hematoma (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Dysphasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Superventricular Tachycardia (SVT) (Cardiac disorders) | 1 (1) | 0 (0)
Intrabdominal hematoma secondary to bike accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Birth by Caesarian Section (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Possible Stroke (Vascular disorders) | 1 (1) | 0 (0)
Fall while intoxicated (Psychiatric disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Left sided weakness (Psychiatric disorders) | 1 (1) | 0 (0)
Fell out of Bed (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ehrlichiosis (Infections and infestations) | 1 (2) | 0 (0)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Induction of Labor (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Septoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Cervical stenosis (Surgical and medical procedures) | 1 (1) | 0 (0)
Laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery with finding of diffuse astrocytoma (Surgical and medical procedures) | 1 (1) | 0 (0)
Cervical myelopathy (Surgical and medical procedures) | 0 (0) | 1 (1)
Sleeve gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cerebral spinal fluid leak (Surgical and medical procedures) | 0 (0) | 1 (1)
Hemicholectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal stenosis (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Med-South Weight Loss Intervention (N=182) | Augmented Usual Care (WW) (N=178)
Hypoglycemia (Metabolism and nutrition disorders) | 14 (19) | 13 (21)
Dizziness (Cardiac disorders) | 22 (30) | 24 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-06-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04302727/Prot_001.pdf
  • Statistical Analysis Plan (2025-06-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT04302727/SAP_002.pdf
  • Informed Consent Form (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT04302727/ICF_000.pdf